CLINICAL TRIAL: NCT05597839
Title: A Phase 1/1b First-In-Human, Multi-Part, Open-Label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of DF9001 as a Monotherapy and in Combination Therapies in Patients With Advanced (Unresectable, Recurrent, or Metastatic) Solid Tumors, and Expansion in Selected Indications
Brief Title: Study of DF9001 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dragonfly Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DF9001-001; KEYNOTE-F92 (Other: Merck); MK-3475-F92 (Other: Merck)
Record Dates: First submitted 2022-10-18; First posted 2022-10-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Adult
Keywords: EGFR; NK Cell; Immunotherapy; Non-Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Renal Cell Carcinoma; pembrolizumab; KEYTRUDA®
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Monotherapy DF9001 Dose Escalation (Experimental): Dose escalation cohorts of DF9001 in sequential ascending order.
  Interventions: Drug: DF9001
- Monotherapy DF9001 Expansion in Head and Neck Squamous Cell Carcinoma (Experimental): Monotherapy expansion cohort enrolling up to 20-40 patients with head and neck squamous cell carcinoma (HNSCC) using the recommended phase 1b dose (REED) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF9001
- Monotherapy DF9001 Expansion in Non-small Cell Lung Cancer (Experimental): Monotherapy expansion cohort enrolling up to 20-40 patients with Non-small cell lung cancer (NSCLC) using the recommended phase 1b dose (REED) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF9001
- Combination Expansion of DF9001 and pembrolizumab in Head and Neck Squamous Cell Carcinoma (Experimental): Combination expansion cohort using DF9001 and a PD-1 checkpoint inhibitor enrolling 20-40 patients with head and neck squamous cell carcinoma (HNSCC) using the recommended phase 1b dose (REED) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF9001; Drug: KEYTRUDA® (pembrolizumab)
- Combination Expansion of DF9001 and pembrolizumab in Renal Cell Carcinoma (Experimental): Combination expansion cohort using DF9001 and a PD-1 checkpoint inhibitor enrolling 20-40 patients with renal cell carcinoma (RCC) using the recommended phase 1b dose (REED) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF9001; Drug: KEYTRUDA® (pembrolizumab)
- Monotherapy DF9001 Expansion in Renal Cell Carcinoma (Experimental): Monotherapy expansion cohort enrolling up to 20-40 patients with renal cell carcinoma (RCC) using the recommended phase 1b dose (REED) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF9001

INTERVENTIONS:
Drug: DF9001 — Immunotherapy agent targeting NK cells.
Drug: KEYTRUDA® (pembrolizumab) — Anti-PD-1 immunotherapy agent
  Arms: Combination Expansion of DF9001 and pembrolizumab in Head and Neck Squamous Cell Carcinoma; Combination Expansion of DF9001 and pembrolizumab in Renal Cell Carcinoma

SUMMARY:
DF9001-001 is a study of a new molecule that targets natural killer (NK) cells and T-cell activation signals to specific receptors on cancer cells. The study will occur in two phases. The first phase will be a dose escalation phase, enrolling patients with various types of solid tumors that express epidermal growth factor receptor (EGFR). The second phase will include a dose expansion using the best dose selected from the first phase of the study. Multiple cohorts will be opened with eligible patients having selected solid tumors (monotherapy and in combination with pembrolizumab).

ELIGIBILITY:
Inclusion Criteria: General (applies to all cohorts)

1. Signed written informed consent.
2. Male or female patients aged ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study entry and an estimated life expectancy of at least 3 months.
4. Adequate hematological function per protocol.
5. Adequate hepatic function per protocol.
6. Adequate renal function per protocol.
7. Participation in the use of contraception during the study, and for 150 days after the last dose of study drug for women of child-bearing potential (WOCBP) and 30 days after the last dose of study drug for male patients, as defined by the Clinical Trial Facilitation Group (CTFG) guidelines.

Inclusion Criteria: Dose Escalation (Monotherapy)

1. Histologically proven locally advanced or metastatic solid tumors of epithelial origin that (1) have squamous NSCLC or HNSCC, (2) has documented EGFR protein expression or EGFR amplification or polysomy in their medical history from previous testing, or (3) test positive for EGFR expression via archival or fresh biopsy tissue prior to study enrollment using a validated immunohistochemistry (IHC) assay.
2. Evidence of objective disease, but participation does not require a measurable lesion.

Inclusion Criteria: Head and Neck Squamous Cell Carcinoma (HNSCC) Expansion Cohorts

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Histologically documented relapsed or metastatic HNSCC. Primary tumor locations include oropharynx, oral cavity, hypopharynx, or larynx. Patients may not have a primary tumor site of nasopharynx (any histology).
3. Patients must have radiographic disease progression while on or after having received both platinum-based or fluoropyrimidine-based chemotherapy and an anti-PD-(L)1 therapy, administered either concurrent or sequentially.
4. Willing and able to provide the most recently available tissue blocks representing tumor biopsy obtained prior to treatment initiation. If recent tissue is not available, then a newly obtained baseline biopsy of an accessible tumor is required. Note that "recent" is defined as no intervening systemic anticancer therapies from the time of the last treatment of the prior therapy until screening for this trial.
5. Willing to undergo on-treatment biopsies, if safe and medically feasible.

Inclusion Criteria: Renal Cell Carcinoma (RCC) Expansion Cohorts

1. Patients must have radiographic progression during treatment or after completing treatment for advanced (recurrent/unresectable/metastatic) disease or be intolerant to prior therapy.
2. Histologically documented relapsed or metastatic RCC that has documented EGFR expression or EGFR gene amplification or polysomy in their medical history from previous testing or test positive for EGFR expression (Section 6.2 EGFR Positivity) via archival (only if a block is available) or fresh biopsy tissue prior to study enrollment using a validated IHC assay. Cytology specimens cannot be used for the purpose of defining EGFR expression to meet eligibility.
3. Patients with clear cell RCC (ccRCC) must have radiographic progression after receipt of one of the following combination regimens as the preceding line of therapy:

   1. PD-1/PD-L1-targeting mAb with or without a VEGFR-TKI.
   2. PD-1-targeting mAb with a CTLA-4 monoclonal.
   3. Patients with non-clear cell RCC (nccRCC) are not required to have received prior therapy in the metastatic setting.
   4. Patients with RCC in general are not required to have received TKI therapy (eg, axitinib, cabozantinib, lenvatinib + everolimus, tivozanib).
4. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
5. Willing and able to provide the most recently available tissue blocks representing tumor biopsy obtained prior to treatment initiation. If recent tissue is not available, then a newly obtained baseline biopsy of an accessible tumor is required. Note that "recent" is defined as no intervening systemic anticancer therapies from the time of the last treatment of the prior therapy until screening for this trial.
6. Willing to undergo on-treatment biopsies, if safe and medically feasible.

Inclusion Criteria: Non-Small Cell Lung Cancer (NSCLC) Expansion Cohorts

1. Histologically confirmed NSCLC meeting stage criteria for stage IIIB, stage IIIC, or stage IV NSCLC disease with or without actionable genomic alterations (AGA) (per the 7th IASLC classification of NSCLC), or recurrent disease.

   1. Patients with squamous NSCLC do not require EGFR testing as part of this study to be eligible.
   2. Non-squamous NSCLC patients who have documented EGFR expression or EGFR gene amplification or polysomy in their medical history from previous testing or test positive for EGFR expression (Section 6.2 EGFR Positivity) via archival (only if a block is available) or fresh biopsy tissue prior to study enrollment using a validated IHC assay.
   3. Patients with stage IIIB or IIIC must be ineligible for local therapies with curative intent (eg, radiotherapy or surgery).
2. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
3. Patients must have recurrent or progressive disease during or after first line combination therapy with checkpoint inhibitors and platinum-based chemotherapy OR must have recurrent or progressive disease within 6 months after completing platinum- based chemotherapy for local disease, including those with actionable genetic alterations. They must not have received any subsequent lines of therapy.
4. Status for actionable mutations (EGFR, ALK, ROS1, RET, etc.) must be known (when testing is available as per country/region standard of care practices); patients with actionable mutations must have received and progressed on, have been intolerant to, or not be a candidate for standard TKIs (as available per country/region standard of care practices).
5. Willing and able to provide the most recently available tissue blocks representing tumor biopsy obtained prior to treatment initiation. If recent tissue is not available, then a newly obtained baseline biopsy of an accessible tumor is required. Note that "recent" is defined as no intervening systemic anticancer therapies from the time of the last treatment of the prior therapy until screening for this trial.
6. Willing to undergo on-treatment biopsies, if safe and medically feasible.

Exclusion Criteria:

1. Patients must not have had chemotherapy, radiotherapy (other than palliative bone- directed radiotherapy, as described in in exclusion criterion #2), or major surgery, or received another investigational agent within 28 days or 5 half-lives of the drug (if known), whichever is shorter, before the start of study treatment.
2. Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids.

   a. Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system (CNS) disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
3. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
4. Concurrent anticancer treatment (eg, cytoreductive therapy, radiotherapy [except for palliative bone-directed radiotherapy, which is not a target lesion], immune therapy, or cytokine therapy [except for erythropoietin]), major surgery (excluding prior diagnostic biopsy), concurrent systemic therapy with steroids or other immunosuppressive agents, or use of any investigational drug within 28 days or 5 half-lives of the drug (if known), whichever is shorter, before the start of study treatment. Short-term administration of systemic steroids (eg, for allergic reactions or the management of irAEs) is allowed. Note: Patients receiving bisphosphonate or denosumab are eligible, provided treatment was initiated at least 14 days before the first dose of DF9001.
5. Previous malignant disease other than the target malignancy to be investigated in this study within the last 3 years. Exceptions (eg, basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ) can be considered on a case-by-case basis, in consultation with the Medical Monitor.
6. Life expectancy of less than 6 months.
7. Receipt of any organ transplantation, including autologous or allogeneic stem-cell transplantation.
8. Significant acute or chronic infections (including historic positive test for human immunodeficiency virus [HIV], or active or latent hepatitis B or active hepatitis C tested during the screening window). If HBsAg is negative and the anti-hepatitis B core antibody is positive, then hepatitis B viral DNA load must be undetectable.
9. Preexisting autoimmune disease (except for patients with vitiligo) needing treatment with systemic immunosuppressive agents for more than 28 days within the last 3 years, or clinically relevant immunodeficiencies (eg, dysgammaglobulinemia or congenital immunodeficiencies). Patients with a history of immune-related endocrinopathies (eg, hypothyroidism, type 1 diabetes mellitus [TIDM], and adrenal insufficiency) that are stable on hormone replacement therapy may be eligible for this study.
10. Patients with a known medical history that may place them at risk of known toxicities of EGFR blockade.

    1. History of or ongoing keratitis, ulcerative keratitis, or corneal perforation.
    2. History of cardiopulmonary arrest unless this was caused by an acute, reversible etiology that is no longer present.
    3. History of or ongoing pulmonary fibrosis or interstitial lung disease.
11. Known severe hypersensitivity reactions to mAbs (≥ Grade 3 of the NCI-CTCAE v5.0), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partly controlled asthma).
12. Persisting toxicity related to prior therapy >Grade 1 NCI-CTCAE v5.0; however, alopecia ≤Grade 2, endocrinopathies ≤Grade 2, and sensory neuropathy ≤ Grade 2 is acceptable.
13. Patients who have received an anti-PD-(L)1 as a previous line of therapy that have experienced either of the following:

    1. a Grade 3 or Grade 4 drug-related toxicity.
    2. a Grade 2 drug-related toxicity that impacted either the lungs, cardiac, or the nervous system, caused by the administration of the anti-PD-(L)1.
14. Received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
15. A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
16. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines are allowed.
17. Pregnancy or lactation in females during the study.
18. Known alcohol or drug abuse.
19. Serious cardiac illness or medical conditions, including but not limited to:

    1. History of New York Heart Association class III or IV heart failure or systolic dysfunction (left ventricular ejection fraction [LVEF] <55%).
    2. High-risk uncontrolled arrhythmias (eg, tachycardia with a heart rate >100/min at rest).
    3. Significant ventricular arrhythmia (ventricular tachycardia) or higher-grade atrioventricular (AV) block (eg, AV-block, second degree AV block Type 2 [Mobitz 2], or third-degree AV-block).
    4. Angina pectoris requiring anti-anginal medication.
    5. Clinically significant valvular heart disease.
    6. Evidence of transmural infarction on electrocardiograms (ECGs).
    7. Poorly controlled hypertension (defined as systolic >160 mm Hg or diastolic >100 mm Hg).
    8. Clinically relevant uncontrolled cardiac risk factors, clinically relevant pulmonary disease, or any clinically relevant medical condition in the opinion of the Investigator that may limit participation in this study.
    9. Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.
20. All other significant diseases (eg, inflammatory bowel disease), which, in the opinion of the Investigator, might impair the patient's ability to participate.
21. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
22. Legal incapacity or limited legal capacity.
23. Incapable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
24. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study treatment (for NSCLC cohorts only).
25. Patients with brain metastases, unless all of the following criteria are met:

    1. CNS lesions are asymptomatic, previously treated and no active therapy is required (ie, no corticosteroids for edema),
    2. Radiologically stable (ie, without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study intervention.
    3. Imaging demonstrates stability of disease 28 days from last treatment for CNS metastases.
26. Active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid).
27. Patients with leptomeningeal disease are excluded.
28. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
29. Active infection requiring systemic therapy.
30. Severe hypersensitivity (≥Grade 3) to pembrolizumab, and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Number, severity, and duration of treatment-related adverse events (TRAEs) according to NCI-CTCAE v5.0. | Screening visit up to 28 days after last treatment on the study.
  To assess the safety of DF9001 by measuring Number of subjects with Treatment-Related Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Number of patients with AEs and TRAEs. | Screening visit up to 28 days after last treatment on the study.
  To assess the safety of DF9001 by measuring Number of subjects with Treatment-Related Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Assessment of number of dose limiting toxicities experienced on study as defined per criteria in the study protocol | First 4 weeks of treatment for each subject.
  To assess the number of adverse events experienced during the study that meet dose limiting toxicity criteria per the study protocol.
Assess Overall Response Rate | Through 90 days after completion of the study, an average of 1 year.
  To assess the Overall Response Rate (ORR) per RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Serum concentrations of DF9001 will be determined at various time points. | From start of treatment up through 7 days after the decision to stop study treatment.
  Concentration vs time of DF9001 will be measured using blood samples taken at various time points on study.
Assess the best overall response (BOR) per RECIST v1.1. | Through 90 days after completion of the study, an average of 1 year.
  To assess Best Overall Response (BOR)
Assess the duration of response (DOR) per RECIST v1.1. | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months.
  To assess Duration of Response (DOR) of DF9001
Assess progression-free survival (PFS) for DF9001 per RECIST v1.1. | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months.
  To assess Progression Free Survival (PFS) for DF9001

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Banner MD Anderson, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UC Irvine Medical Center, Irvine, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Louisville Hospital, Louisville, Kentucky
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - AMR Kansas City, Kansas City, Missouri
  - Rutgers, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UMPC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin